CLINICAL TRIAL: NCT04617418
Title: Using Day-to-day Behavior on Smartphones to Improve Epilepsy Management
Brief Title: Smartphone Behavior and Epilepsy Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stichting Epilepsie Instellingen Nederland (Other)
Collaborators: Leiden University (Other)
Responsible Party: Sponsor
Other Study IDs: SB&EM
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects with refractory focal epilepsy with a seizure frequency: The investigators will include 100 subjects with refractory focal epilepsy with a seizure frequency of at least one per month, and ask them to keep a seizure diary and use the TapCounter app for three months.
  Interventions: Behavioral: Change in touchscreen interactions

INTERVENTIONS:
Behavioral: Change in touchscreen interactions — The investigators will measure the changes in touchscreen interactions using the TapCounter app by QuantActions

SUMMARY:
In this prospective cohort study smartphone behavior surrounding epileptic seizures will be quantified, using a smartphone app, in order to optimize epilepsy evaluation and treatment

DETAILED DESCRIPTION:
Rationale:

The unpredictability of seizures and the unclear behavioral outcomes are major concerns for people with epilepsy and may surface as increased anxiety about independence. This unpredictability is also a true obstacle in capturing and studying seizure-related neurobehavioral alterations themselves. Also, seizures often impact consciousness and thus may go unnoticed. As a result, subjective seizure diaries are unreliable. Continuous smartphone-based monitoring of behavioral output is a fast-emerging topic and proven fruitful in monitoring other neurological disease states. In the field of epilepsy, these tools are yet to be introduced.

Objective:

The investigators hypothesize that quantifying smartphone behavior will help obtain a detailed and objective behavioral map of seizures that can complement existing subjective seizure diaries and thereby improve the way epilepsy treatments are evaluated in daily practice.

Study design:

A multicentre observational prospective cohort study with at least 3 months follow-up.

Study population:

100 subjects with refractory focal epilepsy with a seizure frequency of at least one per month.

Main study parameters/endpoints:

Change in touchscreen interactions (tapping speed, texting speed, apps used, location, sleep-wake cycles) surrounding reported epileptic seizures.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* clinical diagnosis of refractory focal epilepsy meeting ILAE criteria16, 17
* supported by at least one of the following; (1) interictal EEG with epileptiform discharges, (2) epileptogenic lesion on MRI corresponding to the presumed seizure onset zone, or (3) seizure recorded during a video-EEG
* have a seizure frequency of ≥ 1 per month
* only one seizure type, or in case of multiple seizure types only seizures that correspond to one probable onset zone (e.g. focal and focal to bilateral tonic-clonic seizures)
* have daytime seizures (exclusively or both daytime and night-time seizures)
* mentally competent and with no learning disabilities
* able to keep a seizure diary including time and date (as judged by the treating physician)
* have an Android-operating smartphone
* use their phone with at least 5 distinct smartphone apps at a minimum of 5 days a week

Exclusion Criteria:

* not fulfilling the above mentioned inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 subjects with refractory focal epilepsy with a seizure frequency of at least one per month.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in tapping speed surrounding reported epileptic seizures | 3 months
  The tapping speed will be measured using the TapCounter app by QuantActions
Changes in number of apps used surrounding reported epileptic seizures | 3 months
  The number of apps used will be measured using the TapCounter app by QuantActions
Changes in time spent using the smartphone surrounding reported epileptic seizures | 3 months
  The phone usage in hours will be measured using the TapCounter app by QuantActions
Changes in speed of unlocking the smartphone surrounding reported epileptic seizures | 3 months
  The unlocking speed will be measured using the TapCounter app by QuantActions

SECONDARY OUTCOMES:
Recovery after seizure | 3 months
  See how long does it take to behaviorally recover after a seizure, this will be assessed using the TapCounter app and seeing when phone usage before and after the reported seizure are similar again
Comparison of seizures in diaries and seizures in app use | 3 months
  See if reported seizure incidence matches with seizure incidence deducted from smartphone measurements
Subgroup analysis | 3 months
  Analyze differences in behavioural patterns between individuals with different types of epilepsy (e.g. different seizure types or onset zones)

CONTACTS AND LOCATIONS:
Overall Officials: Roland D Thijs, MD PhD, Principal Investigator — Stichting Epilepsie Instellingen Nederland
Locations (4):
- Netherlands (4):
  - Kempenhaeghe, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland, Heemstede, North Holland
  - Maasstad ziekenhuis, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No